CLINICAL TRIAL: NCT05530668
Title: Tolerance and Potential Synergistic Effect of the Combination of Intranasal Esketamine and Non-selective Monoamine Oxidase Inhibitors (MAOIs)
Brief Title: Tolerance and Potential Synergistic Effect of the Combination of Intranasal Esketamine and Non-selective MAOI
Acronym: ESKETAM
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8588
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Depression Anxiety Disorder
Keywords: Depression Disorder; Anxiety Disorder; intranasal esketamine; monoamine oxidase inhibitors (MAOIs); MAOIs; antidepressants; ketamine
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are already recently published data on the tolerability and efficacy of the combination of ketamine and/or esketamine with MAOIs. However, these reports are few and far between, and to our knowledge, there are no data involving intranasal esketamine.

Given the numerous interactions between MAOIs and other antidepressants, and the impossibility of combination, this pharmacological class is neglected. This is despite the fact that MAOIs are the only truly tri-aminergic drugs, that they have unparalleled efficacy in certain forms of resistant apathetic depression, and that new, more dietary permissive forms have appeared on the market. The arrival of antidepressants that can be combined with MAOIs, such as ketamine and esketamine, changes the situation and could offer a new treatment opportunity to many patients in a therapeutic impasse. For these opportunities to become a reality, sharing the clinical experience gained by specialized centers is essential.

ELIGIBILITY:
Inclusion criteria:

* Major subject.
* Having been treated with intranasal esketamine between 01/01/2018 and 01/03/2022.
* Not objecting to the reuse of their data for scientific research purposes.

Exclusion Criteria:

- Subject who has expressed opposition to the reuse of their data for scientific research purposes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject.having been treated with intranasal esketamine between 01/01/2018 and 01/03/2022.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Number of adverse events for each patient | Files analysed retrospectively from January 01, 2018 to March 31, 2022 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de physiologie - Explorations fonctionnelles - CHU de Strasbourg - France, Strasbourg, France

REFERENCES:
- [Derived] Dormegny-Jeanjean LC, Lenoir S, Humbert I, Mainberger OAE, Lozere C, Meyer C, Geny B, Michel B, Foucher JR, de Crespin de Billy C. Cardiovascular Effects of Non-Selective Monoamine Oxidase Inhibitors and Intranasal Esketamine Combination in Depression - A Quasi-Experimental Design with Bayesian Analyses. Pharmacopsychiatry. 2025 Nov;58(6):273-283. doi: 10.1055/a-2590-3469. Epub 2025 Jun 2. PMID 40456292